CLINICAL TRIAL: NCT04250077
Title: SBIR Phase 1: Scalable Digital Delivery of Evidence-based Training for Family to Maximize Treatment Admission Rates of Opioid Use Disorder in Loved Ones-- We The Village Family Support Study
Brief Title: We The Village Family Support Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: We The Village, Inc. (Other)
Collaborators: Public Health Management Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Protocol 1906
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Results first posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-11

CONDITIONS: Community Reinforcement And Family Training; Family Health; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Phase One of this project will develop and refine digital delivery of two modified CRAFT (Community Reinforcement and Family Training) interventions: automated and Group CRAFT protocol (CRAFT-A) and automated CRAFT protocol with live coaching (CRAFT-C) and assess the effectiveness of the adapted CRAFT protocols with WTV's business as usual model of Peer Support Forum (PEER). The goal of the project is to deliver an innovative and effective evidence-based behavioral intervention with consumer technology to an existing and growing online audience.
Who Masked: Outcomes Assessor
Masking Description: The participants will know what group they are in. When we send the data to the statistician for analysis we can code the groups (e.g., 123) and not tell them which is which. This masks (or blinds) him to the condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRAFT-A (Experimental): Participants assigned to the CRAFT-A will have access to a 12-module on-line CRAFT intervention and asked to complete one module weekly for 12 weeks. Modules introduce CRAFT concepts and provide workbooks to assist participants in learning and applying the concepts. The modules include: 1)Introduction to CRAFT; 2) Communication Training; 3) Functional Analysis of Drug Using; 4) Positive Reinforcement; 5) Withdrawing Reinforcement; 6) Allowing Natural Consequences; 7) Problem-solving; 8) Life Enrichment; 9) Suggesting Treatment; 10) Recovery and Relapse; 11) Relationship; and 12) Recap of Skills.
  CRAFT-A participants also attend a weekly 60-minute online group sessions facilitated by a CRAFT-certified coach. During weekly group sessions concepts are briefly reviewed, questions are answered, and skills are practiced through role-plays of common situations.
  Interventions: Behavioral: Community Reinforcement And Family Training (CRAFT)
- CRAFT-C (Experimental): Participants assigned to the CRAFT-C groups will have access to a 12-module on-line CRAFT intervention and asked to complete one module weekly for 12 weeks. Modules introduce CRAFT concepts and provide workbooks to assist participants in learning and applying the concepts. The modules include: 1) Introduction to CRAFT; 2) Communication Training; 3) Functional Analysis of Drug Using; 4) Positive Reinforcement; 5) Withdrawing Reinforcement; 6) Allowing Natural Consequences; 7) Problem-solving; 8) Life Enrichment; 9) Suggesting Treatment; 10) Recovery and Relapse; 11) Relationship; and 12) Recap of Skills.
  CRAFT-C participants attend a weekly 60-minute individualized on-on-one coaching session with a CRAFT certified coach. During weekly individual sessions concepts are briefly reviewed, questions are answered, and skills are practiced through role-plays of common situations. One-on-one sessions involve role-plays that are tailored to the participants' specific circumstances
  Interventions: Behavioral: Community Reinforcement And Family Training (CRAFT)
- PEER (Active Comparator): Participants assigned to the PEER group will participate in an online peer support forum with other CSOs.
  Members of the forum post questions or comments to weekly peer-led discussions and receive responses and feedback from other CSO forum members. Members typically express concerns regarding their IP's wellbeing and ask other members to share any strategies they have employed when dealing with their IPs. Interactions typically, are based either in 12-Step strategies members have learned (usually through Al-Anon or Nar-Anon Family Groups or Family Training Workshops provided by treatment programs) or in CRAFT skills learned (usually from treatment programs or other We The Village members). A staff member from We The Village monitors forum interactions to ensure members are interacting respectfully. This individual also will report any adverse or severe adverse events that members mention online.
  Interventions: Behavioral: We The Village Peer Community Forum

INTERVENTIONS:
Behavioral: Community Reinforcement And Family Training (CRAFT) — Community Reinforcement Approach and Family Training (CRAFT) is a scientifically based intervention designed to help concerned significant others (CSOs) to engage treatment-refusing substance abusers into treatment. This new intervention method was developed with the belief that the CSO can play a powerful role in helping to engage the substance user in treatment. It is often the substance user who reports that family pressure or influence is the reason sought treatment. CSOs benefit by becoming more independent and reducing their depression, anxiety and anger symptoms even if their loved one does not enter treatment.
  CRAFT uses a positive approach versus confrontation, emphasizing learning new skills to cope with old problems. Some components include: how to stay safe, outlining the context in which substance abusing behavior occurs, teaching CSOs how to use positive reinforcers (rewards) and how to let the substance user suffer the natural consequences for their using behavior.
  Arms: CRAFT-A; CRAFT-C
Behavioral: We The Village Peer Community Forum — An online peer support forum with other CSOs. Members of the forum post questions or comments to weekly peer-led discussions and receive responses and feedback from other CSO forum members. Members typically express concerns regarding their IP's wellbeing and ask other members to share any strategies they have employed when dealing with their IPs. Interactions typically, are based either in 12-Step strategies members have learned (usually through Al-Anon or Nar-Anon Family Groups or Family Training Workshops provided by treatment programs) or in CRAFT skills learned (usually from treatment programs or other We The Village members). A staff member from We The Village monitors forum interactions to ensure members are interacting respectfully.
  Arms: PEER

SUMMARY:
The United States is in the midst of an opioid crisis. Over-prescription of opioid analgesic pain relievers contributed to a rapid escalation of use and misuse of these substances across the country. In 2016, more than 2.6 million Americans were diagnosed with opioid use disorder (OUD) and more than 42,000 have died of overdose involving opioids. This death rate is more than any year on record and has quadrupled since 1999 (1,2). Leveraging the potential of available data bases and health IT technologies may help to combat opioid crisis by targeting various aspects of the problem ranging from the prevention of opioid misuse to OUD treatment. NIH through NIDA solicits the research and development of data-driven solutions and services that focus on issues related to opioid use prevention, opioid use, opioid overdose prevention or OUD treatment.

In this project, We The Village, Inc. will address a need to prepare Concerned Significant Others (CSOs) to best use their influence over the trajectory of a loved one's OUD. CSOs are motivated to help, make majority of treatment decisions and payments and have influence over treatment entry and thus, impact the trajectory of an OUD. The project goal is to develop digital delivery of Community Reinforcement And Family Training (CRAFT) methodology, an empirical family behavioral intervention to improve outcomes around treatment entry, family functioning and substance use.

DETAILED DESCRIPTION:
The primary objective of the proposed Phase I work is to determine the feasibility of delivering Community Reinforcement And Family Training (CRAFT) principles via scalable digital coaching methods and determine its efficacy based on measured outcomes.

Technical Objectives 1. Modify the WTV platform to produce a CRAFT-informed automated prototype and protocol for live coaching.

Technical Objectives 2. Test prototype usability and reliability to deliver the protocol, and make any refinements needed.

Technical Objectives 3. Demonstrate prototype efficacy. Testing three digital scenarios: A. Automated CRAFT, B. CRAFT Coach, C. Peer support, the current WTV platform interaction.

As a result, when tested at baseline versus post-intervention, CRAFT conditions (Coach and Automated) are expected to achieve better outcomes than the peer condition in a) treatment entry, b) Concerned Significant Others (CSO) health and wellbeing, c) CSO and identified patient relationship, d) CRAFT adeptness.

Results will substantiate the case for Phase II roll out of the platform at scale, plus commercialization and dissemination through an existing and growing network of partners.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a concerned significant other (CSO) of a loved one with an OUP
* Be 19 years or older
* No substance use disorder
* Has concern about the opioid use of a loved one (IP)
* Plans to be in close contact (phone/face-to-face) with the IP
* The IP is not currently receiving treatment, or the IP is in treatment, but the CSO perceives the IP may benefit from additional treatment (e.g., receiving MAT but the IP may benefit from attending outpatient services, or in residential treatment, but will need to enter outpatient treatment upon discharge).

Exclusion Criteria:

* Does not agree to sign the consent form
* Is not English-speaking
* Is not able to understand the consent form
* Does not have personal access to a smart phone with data or a computer with internet to be able to access the digital platform for the study conditions, quizzes, questionnaires, and follow-up communication
* Reports that they have a drug abuse problem or a history of drug abuse or dependence and that they have not been in recovery for at least 2 years
* Resides outside the United States

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- We the Village, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bischof G, Iwen J, Freyer-Adam J, Rumpf HJ. Efficacy of the Community Reinforcement and Family Training for concerned significant others of treatment-refusing individuals with alcohol dependence: A randomized controlled trial. Drug Alcohol Depend. 2016 Jun 1;163:179-85. doi: 10.1016/j.drugalcdep.2016.04.015. Epub 2016 Apr 19. PMID 27141840
- [Background] Benishek, L. A., Dugosh, K. L., Faranda-Diedrich, T. M., & Kirby, K. C. (2006). Development of the significant other survey: An interview for family members of substance users. American Journal of Family Therapy, 34(1), 33-46.
- [Background] Bresani, E., Kirby, K.C., Meyers, R.J., Case, T., Miller, T.G., Festinger, D.S., Serna, B., & Grasso, S. (2016). The parent's modular toolkit: Development of an online CRAFT program for parents of emerging adults with SUD. Drug and Alcohol Dependence, 156, e27-e28
- [Background] Brigham GS, Slesnick N, Winhusen TM, Lewis DF, Guo X, Somoza E. A randomized pilot clinical trial to evaluate the efficacy of Community Reinforcement and Family Training for Treatment Retention (CRAFT-T) for improving outcomes for patients completing opioid detoxification. Drug Alcohol Depend. 2014 May 1;138:240-3. doi: 10.1016/j.drugalcdep.2014.02.013. Epub 2014 Feb 23. PMID 24656054
- [Background] Center for Behavioral Health Statistics and Quality. (2017.) National Survey on Drug Use and Health: Detailed tables. Rockville, MD: Substance Abuse and Mental Health Services Administration; 2018.
- [Background] Centers for Disease Control (CDC) Multiple Cause of Death 1999-2017 on CDC Wide-ranging Online Data for Epidemiologic Research (CDC WONDER). Atlanta, GA: CDC, National Center for Health Statistics. 2018. Available at http://wonder.cdc.gov.
- [Background] Ghertner, R., & Groves, L. (2018). The opioid crisis and economic opportunity: geographic and economic trends. ASPE Research Brief, 1-22.
- [Background] Hartley, J. (1998). Learning and studying: A research perspective. Florence, KY: Taylor & Frances/Routledge.
- [Background] Hudson CR, Kirby KC, Firely ML, Festinger DS, Marlowe DB. Social adjustment of family members and significant others (FSOs) of drug users. J Subst Abuse Treat. 2002 Oct;23(3):171-81. doi: 10.1016/s0740-5472(02)00245-3. PMID 12392803
- [Background] Kirby KC, Marlowe DB, Festinger DS, Garvey KA, La Monaca V. Community reinforcement training for family and significant others of drug abusers: a unilateral intervention to increase treatment entry of drug users. Drug Alcohol Depend. 1999 Aug 2;56(1):85-96. doi: 10.1016/s0376-8716(99)00022-8. PMID 10462097
- [Background] Kirby KC, Dugosh KL, Benishek LA, Harrington VM. The Significant Other Checklist: measuring the problems experienced by family members of drug users. Addict Behav. 2005 Jan;30(1):29-47. doi: 10.1016/j.addbeh.2004.04.010. PMID 15561447
- [Background] Kirby, K.C., Meyers, K., Carpenedo, C.M., Bresani, E., Dugosh, K.L., Zentgraf, K., & Zaslav, D. (2016). Randomized, controlled trial of CRAFT for parents of treatment-resistant adolescents and young adults: Interim results. Drug and Alcohol Dependence, 156, e112
- [Background] Kirby KC, Benishek LA, Kerwin ME, Dugosh KL, Carpenedo CM, Bresani E, Haugh JA, Washio Y, Meyers RJ. Analyzing components of Community Reinforcement and Family Training (CRAFT): Is treatment entry training sufficient? Psychol Addict Behav. 2017 Nov;31(7):818-827. doi: 10.1037/adb0000306. Epub 2017 Aug 24. PMID 28836796
- [Background] Lovett, L. (2018) Senate passes bill to address opioid crisis, expands telemedicine scope. Mobihealthnews. https://www.mobihealthnews.com/content/senate-passes-bill-address-opioid-crisis-expands-telemedicine- scope?mc_cid=f7c67890d1&mc_eid=3bfb3dd1e7
- [Background] Marlowe DB, Kirby KC, Bonieskie LM, Glass DJ, Dodds LD, Husband SD, Platt JJ, Festinger DS. Assessment of coercive and noncoercive pressures to enter drug abuse treatment. Drug Alcohol Depend. 1996 Oct;42(2):77-84. doi: 10.1016/0376-8716(96)01261-6. PMID 8889406
- [Background] McLellan, A. Thomas Wolfe, B. L., & Meyers, R. J. (2004). Community reinforcement and family training: Getting loved ones sober. In The counselor publication of the National Association of Alcoholism and Drug Abuse Counselors, Vol. 5, No. 3 (pp. 57-60).
- [Background] Meyers RJ, Miller WR, Smith JE, Tonigan JS. A randomized trial of two methods for engaging treatment-refusing drug users through concerned significant others. J Consult Clin Psychol. 2002 Oct;70(5):1182-5. PMID 12362968
- [Background] Meyers, R. J. (2008). Providing a CRAFT book - Get your loved one sober - resulted in treatment entry in greater proportions than seen in twelve-step facilitation control groups. Unpublished raw data.
- [Background] Miller WR, Meyers RJ, Tonigan JS. Engaging the unmotivated in treatment for alcohol problems: a comparison of three strategies for intervention through family members. J Consult Clin Psychol. 1999 Oct;67(5):688-97. doi: 10.1037//0022-006x.67.5.688. PMID 10535235
- [Background] Osilla KC, Kennedy DP, Hunter SB, Maksabedian E. Feasibility of a computer-assisted social network motivational interviewing intervention for substance use and HIV risk behaviors for housing first residents. Addict Sci Clin Pract. 2016 Sep 7;11(1):14. doi: 10.1186/s13722-016-0061-x. PMID 27604543
- [Background] Ray GT, Mertens JR, Weisner C. The excess medical cost and health problems of family members of persons diagnosed with alcohol or drug problems. Med Care. 2007 Feb;45(2):116-22. doi: 10.1097/01.mlr.0000241109.55054.04. PMID 17224773
- [Background] Ray GT, Mertens JR, Weisner C. Family members of people with alcohol or drug dependence: health problems and medical cost compared to family members of people with diabetes and asthma. Addiction. 2009 Feb;104(2):203-14. doi: 10.1111/j.1360-0443.2008.02447.x. PMID 19149814
- [Background] Rhoades H, La Motte-Kerr W, Duan L, Woo D, Rice E, Henwood B, Harris T, Wenzel SL. Social networks and substance use after transitioning into permanentsupportive housing. Drug Alcohol Depend. 2018 Oct 1;191:63-69. doi: 10.1016/j.drugalcdep.2018.06.027. Epub 2018 Jul 29. PMID 30086424
- [Background] Roozen HG, de Waart R, van der Kroft P. Community reinforcement and family training: an effective option to engage treatment-resistant substance-abusing individuals in treatment. Addiction. 2010 Oct;105(10):1729-38. doi: 10.1111/j.1360-0443.2010.03016.x. PMID 20626372
- [Background] Roozen HG, Boulogne JJ, van Tulder MW, van den Brink W, De Jong CA, Kerkhof AJ. A systematic review of the effectiveness of the community reinforcement approach in alcohol, cocaine and opioid addiction. Drug Alcohol Depend. 2004 Apr 9;74(1):1-13. doi: 10.1016/j.drugalcdep.2003.12.006. PMID 15072802
- [Background] Rounsaville, B. J., Carroll, K. M., & Onken, L. S. (2001). A stage model of behavioral therapies research: Getting started and moving on from stage I. Clinical Psychology: Science and Practice, 8(2), 133-142.
- [Background] Scholl L, Seth P, Kariisa M, Wilson N, Baldwin G. Drug and Opioid-Involved Overdose Deaths - United States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2018 Jan 4;67(5152):1419-1427. doi: 10.15585/mmwr.mm675152e1. PMID 30605448
- [Background] Singer, N. (2018) New York Times. Take This App and Call Me in the Morning (March 18) https://www.nytimes.com/2018/03/18/technology/take-this-app-and-call-me-in-the-morning.html
- [Background] Sisson RW, Azrin NH. Family-member involvement to initiate and promote treatment of problem drinkers. J Behav Ther Exp Psychiatry. 1986 Mar;17(1):15-21. doi: 10.1016/0005-7916(86)90005-4. PMID 3700666
- [Background] Slesnick N, Meyers RJ, Meade M, Segelken DH. Bleak and hopeless no more. Engagement Of reluctant substance-abusing runaway youth and their families. J Subst Abuse Treat. 2000 Oct;19(3):215-22. doi: 10.1016/s0740-5472(00)00100-8. PMID 11027890
- [Background] Smyth BP, Barry J, Keenan E, Ducray K. Lapse and relapse following inpatient treatment of opiate dependence. Ir Med J. 2010 Jun;103(6):176-9. PMID 20669601
- [Background] Stanton MD. Getting reluctant substance abusers to engage in treatment/self-help: a review of outcomes and clinical options. J Marital Fam Ther. 2004 Apr;30(2):165-82. doi: 10.1111/j.1752-0606.2004.tb01232.x. PMID 15114946
- [Background] Thomas, E. J., & Santa, C. A. (1982). Unilateral family therapy for alcohol abuse: A working conception. American Journal of Family Therapy, 10(3), 45-58.
- [Background] Thomas, E. J., & Yoshioka, M. R. (1989). Spouse interventive confrontations in unilateral family therapy for alcohol abuse. Social Casework, 70, 340-347.
- [Background] Trudeau JV, Deitz DK, Cook RF. Utilization and cost of behavioral health services: employee characteristics and workplace health promotion. J Behav Health Serv Res. 2002 Feb;29(1):61-74. doi: 10.1007/BF02287832. PMID 11840905
- [Background] Keane H. Facing addiction in America: The Surgeon General's Report on Alcohol, Drugs, and Health U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES, OFFICE OF THE SURGEON GENERAL Washington, DC, USA: U.S. Department of Health and Human Services, 2016 382 pp. online (grey literature): https://addiction.surgeongeneral.gov/. Drug Alcohol Rev. 2018 Feb;37(2):282-283. doi: 10.1111/dar.12578. No abstract available. PMID 29388330
- [Background] van Dommelen-Gonzalez E, Deardorff J, Herd D, Minnis AM. Homies with aspirations and positive peer network ties: associations with reduced frequent substance use among gang-affiliated Latino youth. J Urban Health. 2015 Apr;92(2):322-37. doi: 10.1007/s11524-014-9922-3. PMID 25649980
- [Background] Vice Chairman's Staff of the Joint Economic Committee. (2017). The Numbers Behind the Opioid Crisis: https://www.lee.senate.gov/public/_cache/files/b54a2abb-978d-4bbb-a868-531cdfaeae7a/the-numbers- behind-the-opioid-crisis-final.pdf 2.
- [Background] Ventura AS, Bagley SM. To Improve Substance Use Disorder Prevention, Treatment and Recovery: Engage the Family. J Addict Med. 2017 Sep/Oct;11(5):339-341. doi: 10.1097/ADM.0000000000000331. PMID 28787300
- [Background] Wogan, J.B., (2017). Governing States and Localities. Health and Human Services. For Opioids' Youngest Victims, Is Help Too Little, Too Late? http://www.governing.com/topics/health-human-services/gov-opioid-epidemic- child-welfare.html
- [Derived] Macky JP, Kirby KC, Fitzpatrick BG, Goodwin S, Milnamow M, Kishpaugh J, Lubetkin EJ, Kuecker ML, Bearnot B, Meyers RJ, Handley CJ. Community Reinforcement and Family Training (CRAFT) goes digital: Randomized pilot trial for families of individuals with opioid use problems. Exp Clin Psychopharmacol. 2026 Feb;34(1):78-87. doi: 10.1037/pha0000821. PMID 41538229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began after IRB approval on January 8th 2020 and continued until 45 participants were enrolled on March 16th.
  Online recruitment:
  1. Website callouts, emails, social media posts and 1:1 messages to WTV members.
  2. Outreach to partners who provide services to patients with OUD.
  3. Targeted digital and local advertising efforts.
Pre-assignment Details: Not applicable, people were considered enrolled after baseline interview. 100% of those who completed baseline were assigned to one of the 3 conditions.
Groups:
- CRAFT-C: Participants assigned to the CRAFT-C groups will have access to a 12-module on-line CRAFT intervention and asked to complete one module weekly for 12 weeks. Modules introduce CRAFT concepts and provide workbooks to assist participants in learning and applying the concepts. The modules include: 1) Introduction to CRAFT; 2) Communication Training; 3) Functional Analysis of Drug Using; 4) Positive Reinforcement; 5) Withdrawing Reinforcement; 6) Allowing Natural Consequences; 7) Problem-solving; 8) Life Enrichment; 9) Suggesting Treatment; 10) Recovery and Relapse; 11) Relationship; and 12) Recap of Skills.
  CRAFT-C participants attend a weekly 60-minute individualized on-on-one coaching session with a CRAFT certified coach. During weekly individual sessions concepts are briefly reviewed, questions are answered, and skills are practiced through role-plays of common situations. One-on-one sessions involve role-plays that are tailored to the participants' specific circumstances
  Community R
- PEER: Participants assigned to the PEER group will participate in an online peer support forum with other CSOs.
  Members of the forum post questions or comments to weekly peer-led discussions and receive responses and feedback from other CSO forum members. Members typically express concerns regarding their IP's wellbeing and ask other members to share any strategies they have employed when dealing with their IPs. Interactions typically, are based either in 12-Step strategies members have learned (usually through Al-Anon or Nar-Anon Family Groups or Family Training Workshops provided by treatment programs) or in CRAFT skills learned (usually from treatment programs or other We The Village members). A staff member from We The Village monitors forum interactions to ensure members are interacting respectfully. This individual also will report any adverse or severe adverse events that members mention online.
  We The Village Peer Community Forum: An online peer support forum with other CSOs.
  M
Period: Overall Study
Arm/Group | CRAFT-A | CRAFT-C | PEER
Started | 15 | 15 | 15
Completed | 13 | 11 | 15
Not Completed | 2 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRAFT-A | CRAFT-C | PEER | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] — Self administered online tool, continuous variable - how old are you. Population: Stratified random assignment was conducted to ensure equal number of enrolled participants across conditions.
  Years | 38.3 (10.6) | 45.2 (12.5) | 46.3 (11.2) | 43.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Self administered online tool. Categorical measure for gender. Population: Stratified random assignment was conducted to ensure equal number of enrolled participants across conditions.
  Participants
    Female | 14 | 15 | 13 | 42
    Male | 1 | 0 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self administered online tool, categorical variable - what is your ethnicity? Population: Stratified random assignment was conducted to ensure equal number of enrolled participants across conditions.
  Participants
    Hispanic or Latino | 2 | 0 | 0 | 2
    Not Hispanic or Latino | 12 | 14 | 15 | 41
    Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self administered online tool, categorical variable - what is your race, check all that apply. Population: Stratified random assignment was conducted to ensure equal number of enrolled participants across conditions.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 15 | 13 | 14 | 42
    More than one race | 0 | 2 | 1 | 3
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45
IP current treatment status for OUD [Count of Participants; unit: Participants] — Self administered online tool, categorical variable - is your loved one currently engaged in treatment for their opioid use problem.
  Participants
    Yes | 6 | 6 | 6 | 18
    No | 7 | 9 | 9 | 25
    Don't know | 2 | 0 | 0 | 2
Relationship Happiness Scale [Mean (Standard Deviation); unit: units on a scale] — 10-item standardized scale used to measure current happiness in a person's relationship in 9 domains and overall, on a scale from 1-10. Global score is calculated by adding scores from 10 items. Minimum possible score is 10 and maximum is 100. Higher scores reflect greater Relationship Happiness. Self-report, electronic data collection method. Population: Per IRB approval and requirements, survey questions were optional and so some participants opted out of responding to particular questions.
  units on a scale
    number analyzed (Participants) | 11 | 10 | 12 | 33
    (all) | 26.15 (10.90) | 23.45 (15.47) | 35.43 (19.62) | 28.789473684210 (16.309768080835)
Profile of Mood State (POMS) - Short Form [Mean (Standard Deviation); unit: units on a scale] — 37-item standardized scale used to measure mood on a scale from 1-5 across 6 subscales (tension, depression, anger, vigor, fatigue, confusion) with a total mood disturbance (TMD) score calculated by adding scores from the tension (6 items), depression (8 items), anger (7 items), fatigue (5 items), and confusion (5 items) subscales, then subtracting the score form the vigor (6 items) subscale. Minimum TMD possible score is 1 and maximum is 149. Higher scores reflect greater mood disturbance. Self-report, electronic data collection method. Population: Per IRB approval and requirements, survey questions were optional and so some participants opted out of responding to particular questions.
  units on a scale
    number analyzed (Participants) | 10 | 10 | 12 | 32
    (all) | 99.46153846 (25.76695359) | 84.63636364 (29.26182745) | 79.6 (34.91990836) | 87.641025641025 (30.986828423742)
CRAFT Knowledge Scale [Mean (Standard Deviation); unit: units on a scale] — Adapted family training survey for OUD population. 10 scenarios, multiple choice with only one correct answer per scenario. Knowledge score calculated by adding the number of correct answers. Minimum score is 0 and maximum is 10. Higher score reflects higher knowledge. Self-report, electronic data collection method. Population: Per IRB approval and requirements, survey questions were optional and so some participants opted out of responding to particular questions.
  units on a scale
    number analyzed (Participants) | 13 | 11 | 15 | 39
    (all) | 4.230769231 (2.241794153) | 4.090909091 (1.375103302) | 4.133333333 (1.552264091) | 4.1538461538461 (1.7250242033155)
SF-12 Physical Health Subscale [Mean (Standard Deviation); unit: units on a scale] — 7-item subscale of the SF-12 assesses impact of physical health on an individual's daily life. Scored using norm-based methods and transformed so that the scale has a mean of 50 and a s.d. of 10 in the general US population so that all scores above and below 50 are above and below the average with each point representing a difference of 1/10th of a standard deviation.
  Self-report, electronic data collection method. Population: Per IRB approval and requirements, survey questions were optional and so some participants opted out of responding to particular questions.
  units on a scale
    number analyzed (Participants) | 11 | 10 | 12 | 33
    (all) | 48.26037769 (6.807966535) | 46.73253 (10.49979736) | 46.96861067 (12.19914184) | 47.332612820512 (9.9462284409113)
SF-12 Mental Health Subscale [Mean (Standard Deviation); unit: units on a scale] — 5-item subscale of the SF-12 assesses impact of mental health on an individual's daily life. Scored using norm-based methods and transformed so that the scale has a mean of 50 and a s.d. of 10 in the general US population so that all scores above and below 50 are above and below the average with each point representing a difference of 1/10th of a standard deviation.
  Self-report, electronic data collection method. Population: Per IRB approval and requirements, survey questions were optional and so some participants opted out of responding to particular questions.
  units on a scale
    number analyzed (Participants) | 11 | 10 | 12 | 33
    (all) | 31.31094692 (4.814387593) | 34.50071182 (6.312676025) | 33.94517267 (6.266345365) | 33.223787948717 (5.8482705701241)
SAS-SR [Mean (Standard Deviation); unit: units on a scale] — Standardized scale to assess individual's level of satisfaction in their role performance over the past two weeks key life areas. We used subscales representing three areas of work functioning: Work (6 items), Housework (6 items), School (6 items). Each item is scored on a 1-5 scale. Lower scores equal higher satisfaction in their role performance. Minimum score for each subscale is 6 and maximum is 30. Self-report, electronic data collection method. Population: Per IRB approval and requirements, survey questions were optional and so some participants opted out of responding to particular questions. Also, for this measure, it only applied to those who held a paid working position.
  units on a scale
    number analyzed (Participants) | 6 | 8 | 7 | 21
    (all) | 11.57142857 (2.935821456) | 10.2 (3.425395354) | 11.25 (2.815771906) | 10.92 (3.0402850743529)
MAT Status [Count of Participants; unit: Participants] — This is a frequency count of the number of participants who reported that their loved one was currently engaged in treatment for their opioid use problem Population: Per IRB approval and requirements, survey questions were optional and so some participants opted out of responding to particular questions.
  Participants
    number analyzed (Participants) | 13 | 11 | 15 | 39
    (all) | 6 | 4 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Treatment Entry: IP Treatment Status
Description: Participants reported whether their loved one had attended any treatment for their opioid problem since the last assessment by answering 8 questions regarding participation in treatment (e.g., detox, any treatment, new treatment, MAT, new MAT, counseling, support group, and other group). Reports of new treatment, new MAT, and treatment at the follow-up assessment which were not reported at baseline were categorized as treatment entry. In addition, entry into WTV recovery coaching, WTV family coaching, or reports of treatment entry to WTV staff were categorized as treatment entry. Outcome was the proportion of participants reporting that their loved one entered new treatment.
Time Frame: 3-month post study
Population: CRAFT-A: 13/15 final surveys collected, could not reach 2 of the participants. CRAFT-C: 11/15 final surveys collected, could not reach 3 of the participants, 1 participant removed themselves.
  PEER: All participants completed final surveys.
Measure: Number; unit: count of participants
Groups:
- CRAFT-A: Participants assigned to the CRAFT-A will have access to a 12-module on-line CRAFT intervention and asked to complete one module weekly for 12 weeks. Modules introduce CRAFT concepts and provide workbooks to assist participants in learning and applying the concepts. The modules include: 1)Introduction to CRAFT; 2) Communication Training; 3) Functional Analysis of Drug Using; 4) Positive Reinforcement; 5) Withdrawing Reinforcement; 6) Allowing Natural Consequences; 7) Problem-solving; 8) Life Enrichment; 9) Suggesting Treatment; 10) Recovery and Relapse; 11) Relationship; and 12) Recap of Skills.
  CRAFT-A participants also attend a weekly 60-minute online group sessions facilitated by a CRAFT-certified coach. During weekly group sessions concepts are briefly reviewed, questions are answered, and skills are practiced through role-plays of common situations.
  Community Reinforcement And Family Training (CRAFT): Community Reinforcement Approach and Family Training (CRAFT)
- CRAFT-C: Participants assigned to the CRAFT-C groups will have access to a 12-module on-line CRAFT intervention and asked to complete one module weekly for 12 weeks. Modules introduce CRAFT concepts and provide workbooks to assist participants in learning and applying the concepts. The modules include: 1) Introduction to CRAFT; 2) Communication Training; 3) Functional Analysis of Drug Using; 4) Positive Reinforcement; 5) Withdrawing Reinforcement; 6) Allowing Natural Consequences; 7) Problem-solving; 8) Life Enrichment; 9) Suggesting Treatment; 10) Recovery and Relapse; 11) Relationship; and 12) Recap of Skills.
  CRAFT-C participants attend a weekly 60-minute individualized on-on-one coaching session with a CRAFT certified coach. During weekly individual sessions concepts are briefly reviewed, questions are answered, and skills are practiced through role-plays of common situations. One-on-one sessions involve role-plays that are tailored to the participants' specific circumstances.
  Community Reinforcement And Family Training (CRAFT): Community Reinforcement Approach and Family Training (CRAFT)
- PEER: Participants assigned to the PEER group will participate in an online peer support forum with other CSOs.
  Members of the forum post questions or comments to weekly peer-led discussions and receive responses and feedback from other CSO forum members. Members typically express concerns regarding their IP's wellbeing and ask other members to share any strategies they have employed when dealing with their IPs. Interactions typically, are based either in 12-Step strategies members have learned (usually through Al-Anon or Nar-Anon Family Groups or Family Training Workshops provided by treatment programs) or in CRAFT skills learned (usually from treatment programs or other We The Village members). A staff member from We The Village monitors forum interactions to ensure members are interacting respectfully. This individual also will report any adverse or severe adverse events that members mention online.
  We The Village Peer Community Forum: An online peer support forum with other CSOs.
Arm/Group | CRAFT-A | CRAFT-C | PEER
Number analyzed (Participants) | 13 | 11 | 15
count of participants | 10 | 8 | 6
Statistical Analysis 1: Comparison: CRAFT-A vs PEER; Test type: Superiority; p = 0.02578184, Agresti Caffo proportion comparison; proportion = 0.36923076, 95% CI 2-sided [-0.0021812 to 0.64531855], Standard Error of Mean 0.16518156

2. Secondary Outcome: Relationship Happiness: Relationship Happiness Scale
Description: Global score from the 10-item scale was calculated by adding scores (1-10) from 10 items. Minimum possible score was 10 and maximum was 100. Higher scores reflect greater Relationship Happiness.
Time Frame: 3-month post study
Population: CRAFT-A: 11/15 final surveys collected, could not reach 2 of the participants and 2 chose not to respond to this measure.
  CRAFT-C: 10/15 final surveys collected, could not reach 3 of the participants, 1 participant removed themselves, and 1 chose not to respond to this measure.
  PEER: 12/15 All participants completed final surveys but 3 chose not to respond to this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRAFT-A | CRAFT-C | PEER
Number analyzed (Participants) | 11 | 10 | 12
units on a scale | 21.54545455 (4.993384053) | 23.3 (6.645048282) | 1.5 (5.761023688)
Statistical Analysis 1: Comparison: CRAFT-A vs PEER; Test type: Superiority; p = 0.00787297, t-test, 1 sided; Mean Difference (Net) = 20.0454545, 95% CI 2-sided [4.18213496 to 35.9087741], Standard Error of Mean 7.62386242

3. Secondary Outcome: CSO Health and Wellbeing: Profile of Mood State (POMS) - Short Form
Description: Total mood disturbance (TMD) score calculated by adding scores (1-5) from the tension (6 items), depression (8 items), anger (7 items), fatigue (5 items), and confusion (5 items) subscales, then subtracting the score form the vigor (6 items) subscale. Minimum TMD possible score was 1 and maximum was 149. Higher scores reflect greater mood disturbance.
Time Frame: 3-month post study
Population: CRAFT-A: 10/15 final surveys collected, could not reach 2 of the participants, 3 chose not to respond to this measure.
  CRAFT-C: 10/15 final surveys collected, could not reach 3 of the participants, 1 participant removed themselves, 1 chose not to respond to this measure.
  PEER: 12/15 All participants completed final surveys, 3 chose not to respond to this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRAFT-A | CRAFT-C | PEER
Number analyzed (Participants) | 10 | 10 | 12
units on a scale | -43.1 (14.26218777) | -28.8 (11.44241622) | -3.916666667 (6.862787592)
Statistical Analysis 1: Comparison: CRAFT-A vs PEER; Test type: Superiority; p = 0.01387108, t-test, 1 sided; Mean Difference (Net) = -39.183333, 95% CI 2-sided [-73.356073 to -5.0105927], Standard Error of Mean 15.8274398

4. Secondary Outcome: CSO Health and Wellbeing: SF-12 Physical Health Subscale
Description: The 7-item scale was transformed so that is had a mean of 50 and a s.d. of 10 in the general US population. Scores above and below 50 are above and below the average with each point representing a difference of 1/10th of a standard deviation.
Time Frame: 3-month post study
Population: CRAFT-A: 11/15 final surveys collected, could not reach 2 of the participants, 2 chose not to respond to this measure.
  CRAFT-C: 10/15 final surveys collected, could not reach 3 of the participants, 1 participant removed themselves, 2 chose not to respond to this measure.
  PEER: 12/15 All participants completed final surveys, 3 chose not to respond to this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRAFT-A | CRAFT-C | PEER
Number analyzed (Participants) | 11 | 10 | 12
units on a scale | 5.309448182 (2.481191221) | 0.192893 (3.195979184) | -3.127840833 (2.150194321)
Statistical Analysis 1: Comparison: CRAFT-A vs PEER; Test type: Superiority; p = 0.00908118, t-test, 1 sided; Mean Difference (Net) = 8.43728901, 95% CI 2-sided [1.59437702 to 15.2802010], Standard Error of Mean 3.28323704

5. Secondary Outcome: CSO Health and Wellbeing: SF-12 Mental Health Subscale
Description: The 5-item scale was transformed so that is had a mean of 50 and a s.d. of 10 in the general US population. Scores above and below 50 are above and below the average with each point representing a difference of 1/10th of a standard deviation.
Time Frame: 3-month post study
Population: CRAFT-A: 11/15 final surveys collected, could not reach 2 of the participants, 2 chose not to respond to this measure.
  CRAFT-C: 10/15 final surveys collected, could not reach 3 of the participants, 1 participant removed themselves, 1 chose not to respond to this measure.
  PEER: 12/15 All participants completed final surveys, 3 chose not to respond to this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CRAFT-C: Participants assigned to the CRAFT-C groups will have access to a 12-module on-line CRAFT intervention and asked to complete one module weekly for 12 weeks. Modules introduce CRAFT concepts and provide workbooks to assist participants in learning and applying the concepts. The modules include: 1) Introduction to CRAFT; 2) Communication Training; 3) Functional Analysis of Drug Using; 4) Positive Reinforcement; 5) Withdrawing Reinforcement; 6) Allowing Natural Consequences; 7) Problem-solving; 8) Life Enrichment; 9) Suggesting Treatment; 10) Recovery and Relapse; 11) Relationship; and 12) Recap of Skills.
  CRAFT-C participants attend a weekly 60-minute individualized on-on-one coaching session with a CRAFT certified coach. During weekly individual sessions concepts are briefly reviewed, questions are answered, and skills are practiced through role-plays of common situations. One-on-one sessions involve role-plays that are tailored to the participants' specific circumstances
  Community Reinforcement And Family Training (CRAFT): Community Reinforcement Approach and Family Training (CRAFT)
Arm/Group | CRAFT-A | CRAFT-C | PEER
Number analyzed (Participants) | 11 | 10 | 12
units on a scale | 0.23875 (2.415675325) | 0.782613 (2.49361256) | -1.238238333 (2.783141683)
Statistical Analysis 1: Comparison: CRAFT-A vs PEER; Test type: Superiority; p = 0.34633293, t-test, 1 sided; Mean Difference (Net) = 1.47698833, 95% CI 2-sided [-6.1910435 to 9.14502026], Standard Error of Mean 3.68529034

6. Secondary Outcome: CSO Health and Wellbeing: SAS-SR Work Subscale
Description: Social Adjustment Scale, Self-Report. Standardized scale to assess individual's level of satisfaction in their role performance over the past two weeks key life areas. We used subscales representing the work, housework, and school areas of functioning. Each subscale consisted of 6 items scored on a 1-5 scale. A subscale adjustment score was obtained by summing the scores of all the items and dividing by the number of items actually answered. Thus, each subscale summary score had a minimum score of 1 and a maximum score of 5. Lower scores indicate higher satisfaction in their role performance.
Time Frame: 3-month post study
Population: CRAFT-A: 7/15 final surveys collected, could not reach 2 of the participants, 6 chose not to respond to this measure or it did not apply.
  CRAFT-C: 8/15 final surveys collected, could not reach 3 of the participants, 1 participant removed themselves, 3 chose not to respond to this measure or it did not apply.
  PEER: 9/15 All participants completed final surveys, 6 chose not to respond to this measure or it did not apply.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRAFT-A | CRAFT-C | PEER
Number analyzed (Participants) | 7 | 8 | 9
units on a scale | 0.5714285714 (0.2020305089) | -0.875 (0.6105471785) | 0.2222222222 (0.5211573066)
Statistical Analysis 1: Comparison: CRAFT-A vs PEER; Test type: Superiority; p = 0.57872623, t-test, 1 sided; Mean Difference (Final Values) = -0.4285714, 95% CI 2-sided [-5.4078121 to 4.55066924], Standard Error of Mean 2.07315199

7. Secondary Outcome: CRAFT Knowledge: CRAFT Knowledge Scale
Description: Knowledge score calculated by adding the number of correct multiple-choice answers to 10 scenarios. Minimum score was 0 and maximum was 10. Higher scores reflect greater knowledge.
Time Frame: 3-month post study
Population: CRAFT-A: 13/15 final surveys collected, could not reach 2 of the participants. CRAFT-C: 11/15 final surveys collected, could not reach 3 of the participants, 1 participant removed themselves.
  PEER: 15/15 All participants completed final surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CRAFT-A: Participants assigned to the CRAFT-A will have access to a 12-module on-line CRAFT intervention and asked to complete one module weekly for 12 weeks. Modules introduce CRAFT concepts and provide workbooks to assist participants in learning and applying the concepts. The modules include: 1)Introduction to CRAFT; 2) Communication Training; 3) Functional Analysis of Drug Using; 4) Positive Reinforcement; 5) Withdrawing Reinforcement; 6) Allowing Natural Consequences; 7) Problem-solving; 8) Life Enrichment; 9) Suggesting Treatment; 10) Recovery and Relapse; 11) Relationship; and 12) Recap of Skills.
  CRAFT-A participants also attend a weekly 60-minute online group sessions facilitated by a CRAFT-certified coach. During weekly group sessions concepts are briefly reviewed, questions are answered, and skills are practiced through role-plays of common situations.
  Community Reinforcement And Family Training (CRAFT): Community Reinforcement Approach and Family Training (CRAFT
Arm/Group | CRAFT-A | CRAFT-C | PEER
Number analyzed (Participants) | 13 | 11 | 15
units on a scale | 1.692307692 (0.4985185153) | 1.454545455 (0.8131156282) | 0.4 (0.6458659746)
Statistical Analysis 1: Comparison: CRAFT-A vs PEER; Test type: Superiority; p = 0.06283641, t-test, 1 sided; Median Difference (Net) = 1.29230769, 95% CI 2-sided [-0.3873203 to 2.97193574], Standard Error of Mean 0.81588207

8. Secondary Outcome: MAT
Description: Participants reported whether their loved one had attended any treatment for their opioid problem since the last assessment by answering 8 questions regarding participation in treatment. Reports of new MAT and MAT at the follow-up assessment which was not reported at baseline were categorized as new MAT. In addition, reports of MAT entry to WTV staff were included. Outcome was the proportion of participants reporting that their loved one entered MAT. This differs from Outcome Measure 1 in that Outcome Measure 1 included drug-free and medication-assisted treatments of any type, while this measure included only MAT.
Time Frame: 3-month post study
Measure: Count of Participants; unit: Participants
Arm/Group | CRAFT-A | CRAFT-C | PEER
Number analyzed (Participants) | 13 | 11 | 15
Participants | 5 | 3 | 4
Statistical Analysis 1: Comparison: CRAFT-A vs PEER; Test type: Superiority; p = 0.26422281, Agresti Caffo proportion comparison; proportion = 0.11794871, 95% CI 2-sided [-0.2233244 to 0.43508919], Standard Error of Mean 0.16796576

ADVERSE EVENTS:
Time Frame: Participants were assessed at 3 and 6 months post baseline. Adverse event reporting could occur at these assessments or as a function of spontaneous reports occurring during weekly sessions in the CRAFT groups.
Arm/Group | CRAFT-A | CRAFT-C | PEER
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT04250077/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT04250077/SAP_001.pdf
  • Informed Consent Form (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT04250077/ICF_002.pdf